CLINICAL TRIAL: NCT02050204
Title: Evaluating the Health Benefits of Workplace Policies and Practices - Phase II
Acronym: WFHS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH); Office of Behavioral and Social Sciences Research (OBSSR) (NIH); National Institute for Occupational Safety and Health (NIOSH/CDC) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Lisa Berkman, Professor, Harvard School of Public Health (HSPH)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: P16633; U01AG027669 (NIH); U01HD051218 (NIH); U01HD051256 (NIH); U01HD051276 (NIH); U01HD051217 (NIH); R01HL107240 (NIH); U01OH008788 (NIH); U01HD059773 (NIH)
Record Dates: First submitted 2014-01-28; First posted 2014-01-30 (Estimated); Last update posted 2017-12-15 (Actual); Status verified 2017-12

CONDITIONS: Focus of Study: Work Conditions
Keywords: work to family conflict; supervisor support; long work hours; cardiometabolic risk; sleep duration; insomnia symptoms
MeSH Terms: interventions — Methods

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- LEEF Industry only: Intervention (Experimental): Customized to the "Leef" (alias) workplace: A 3-month structural and social change process designed to increase employee control over work time and family supportive supervisory behaviors.
  Interventions: Behavioral: Intervention
- LEEF Industry only: Usual Practice (No Intervention): Continued work conditions and practice as "Usual Practice" in that workplace
- TOMO Industry only: Intervention (Experimental): Customized to the "Tomo" (alias) workplace: A 3-month structural and social change process designed to increase employee control over work time and family supportive supervisory behaviors.
  Interventions: Behavioral: Intervention
- TOMO Industry only: Usual Practice (No Intervention): Continued work conditions and practice as "Usual Practice" in that workplace

INTERVENTIONS:
Behavioral: Intervention — The intervention was a 3-month structural and social change process designed to increase employee control over work time and family supportive supervisory behaviors (Kossek et al., in press). The change process was an integration of two previously evaluated interventions (Hammer et al., 2011; Kelly et al., 2011). A facilitator led 8 hrs of participatory sessions to transition employees from a time-based to a results-based work culture. Supervisors participated in all change activities plus 4hrs of training in supportive supervision. Training in family supportive supervision was implemented with behavioral computer-based training (cTRAIN, NWeta, Lake Oswego, OR) followed by 2 rounds of goal-setting and behavioral self-monitoring using an iPod Touch (Habitrack, OHSU, Portland, OR).
  Arms: LEEF Industry only: Intervention; TOMO Industry only: Intervention

SUMMARY:
Although the prevalence of "family-friendly" policies in US workplaces has increased dramatically, few have been studied using scientifically sound designs. To address this, the NIH and CDC formed the Work, Family, and Health Network (WFHN). During Phase 1, the WFHN designed and conducted multiple pilot and feasibility studies. For Phase 2, the WFHN implemented an innovative intervention based on Phase I pilot studies that is designed to increase family-supportive supervisor behaviors and employee control over work, and to evaluate the intervention using a group randomized experimental design. Customized interventions were performed separately in workplaces of two separate corporate partners.

DETAILED DESCRIPTION:
Although the prevalence of "family-friendly" policies in US workplaces has increased dramatically in recent years, few have been studied using scientifically sound designs. To address this critical gap, the NIH and CDC formed the Work, Family, and Health Network (WFHN). During Phase 1, the WFHN designed and conducted multiple pilot and feasibility studies.

For Phase 2, the WFHN implemented an innovative intervention based on Phase 1 pilot studies that is designed to increase family-supportive supervisor behaviors and employee control over work, and to evaluate the intervention using a group randomized experimental design. The goal of the study is to assess the effects of a workplace intervention designed to reduce work-family conflict, and thereby improve the health and well being of employees. The study intervention is grounded in theory from multiple disciplines and supported by findings from pilot/feasibility studies. The study seeks to inform the implementation of evidence-based, family-friendly policies, and thereby improving the health and well-being of employees and their families nationwide.

The investigators assess the efficacy of the intervention via two independent, group-randomized field experiments, one at each of two employers representing different industries, referred to by alias as "LEEF" and "TOMO". LEEF is an extended care (nursing home) company and facilities were excluded if they were in very isolated settings, if there were fewer than 30 direct patient-care employees, or if facilities were recently acquired. TOMO is an Information Technology company. Within each industry partner, worksites of 50-120 employees each were randomly assigned to intervention or usual practice conditions. All employee and supervisor participants were assessed at baseline and at 6-, 12-, and 18-months post baseline, including survey interviews and health assessments.

Primary health outcomes were comprised of a cardiometabolic risk score using selected biomarkers and sleep duration and quality objectively measured using wrist actigraphy. These primary health outcomes were independently assessed as change from baseline to the 12-month wave, and separately in the two industries.

ELIGIBILITY:
Inclusion Criteria:

* LEEF: employees and supervisors with at least 22 weekly hours of direct patient care work in selected facilities
* TOMO: employees and supervisors located in the two data collection cities

Exclusion Criteria:

* LEEF: nightwork schedule
* TOMO: independent contractor classification

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2753 (Actual)
Dates: Start 2009-09; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Change in total sleep time | baseline to one year later
  Average 24 hour total sleep time as assessed by ~1 week of actigraphy
change in wake after sleep onset | baseline to one year later
  Amount of nightime wake after sleep onset as assessed by ~1 week of actigraphy
change in cardiometabolic risk score | baseline to one year later
  The cardiometabolic risk score was created based on modifiable risk factors using an independently validated CVD risk score developed from the Framingham offspring study; including BMI, blood pressure, HbA1C, cholesterol, and tobacco consumption.

SECONDARY OUTCOMES:
change in sleep insufficiency | baseline to one year later
  Sleep insufficiency was assessed by the following question: How often during the past 4 weeks did you get enough sleep to feel rested upon waking up? Would you say never, rarely, sometimes, often, or very often?
  YES - NEVER/RARELY
  NO - SOMETIMES OFTEN VERY OFTEN
change in insomnia symptoms | baseline to one year later
  Insomnia symptoms were assessed by the following question: During the past 4 weeks, how often did you wake up in the middle of the night or early morning? (Would you say never, less than once a week, once or twice a week, or three or more times a week?)
  YES - THREE OR MORE TIMES A WEEK
  NO - NEVER/LESS THAN ONCE A WEEK/ONCE OR TWICE A WEEK

CONTACTS AND LOCATIONS:
Overall Officials: Lisa F Berkman, PhD, Principal Investigator — Harvard School of Public Health (HSPH); Orfeu M Buxton, PhD, Principal Investigator — Brigham and Women's Hospital; Harvard Medical School; Harvard School of Public Health; Pennsylvania State University
Locations (1):
- Harvard School of Public Health, Cambridge, Massachusetts, United States

REFERENCES:
- [Background] Okechukwu CA, Souza K, Davis KD, de Castro AB. Discrimination, harassment, abuse, and bullying in the workplace: contribution of workplace injustice to occupational health disparities. Am J Ind Med. 2014 May;57(5):573-86. doi: 10.1002/ajim.22221. Epub 2013 Jun 27. PMID 23813664
- [Background] Hammer LB, Ernst Kossek E, Bodner T, Crain T. Measurement development and validation of the Family Supportive Supervisor Behavior Short-Form (FSSB-SF). J Occup Health Psychol. 2013 Jul;18(3):285-96. doi: 10.1037/a0032612. Epub 2013 Jun 3. PMID 23730803
- [Background] Liu S, Rovine MJ, Klein LC, Almeida DM. Synchrony of diurnal cortisol pattern in couples. J Fam Psychol. 2013 Aug;27(4):579-88. doi: 10.1037/a0033735. PMID 23978320
- [Background] Cunningham TJ, Seeman TE, Kawachi I, Gortmaker SL, Jacobs DR, Kiefe CI, Berkman LF. Racial/ethnic and gender differences in the association between self-reported experiences of racial/ethnic discrimination and inflammation in the CARDIA cohort of 4 US communities. Soc Sci Med. 2012 Sep;75(5):922-31. doi: 10.1016/j.socscimed.2012.04.027. Epub 2012 May 23. PMID 22682683
- [Background] O'Donnell EM, Berkman LF, Subramanian SV. Manager support for work-family issues and its impact on employee-reported pain in the extended care setting. J Occup Environ Med. 2012 Sep;54(9):1142-9. doi: 10.1097/JOM.0b013e3182554af4. PMID 22892547
- [Background] Nelson CC, Li Y, Sorensen G, Berkman LF. Assessing the relationship between work-family conflict and smoking. Am J Public Health. 2012 Sep;102(9):1767-72. doi: 10.2105/AJPH.2011.300413. Epub 2012 Jun 21. PMID 22720765
- [Background] Hurtado DA, Sabbath EL, Ertel KA, Buxton OM, Berkman LF. Racial disparities in job strain among American and immigrant long-term care workers. Int Nurs Rev. 2012 Jun;59(2):237-44. doi: 10.1111/j.1466-7657.2011.00948.x. Epub 2011 Dec 7. PMID 22591096
- [Background] Sembajwe G, Wahrendorf M, Siegrist J, Sitta R, Zins M, Goldberg M, Berkman L. Effects of job strain on fatigue: cross-sectional and prospective views of the job content questionnaire and effort--reward imbalance in the GAZEL cohort. Occup Environ Med. 2012 Jun;69(6):377-84. doi: 10.1136/oem.2010.063503. Epub 2011 Aug 17. PMID 21849345
- [Background] Wahrendorf M, Sembajwe G, Zins M, Berkman L, Goldberg M, Siegrist J. Long-term effects of psychosocial work stress in midlife on health functioning after labor market exit--results from the GAZEL study. J Gerontol B Psychol Sci Soc Sci. 2012 Jul;67(4):471-80. doi: 10.1093/geronb/gbs045. Epub 2012 Apr 29. PMID 22546992
- [Background] Okechukwu CA, El Ayadi AM, Tamers SL, Sabbath EL, Berkman L. Household food insufficiency, financial strain, work-family spillover, and depressive symptoms in the working class: the Work, Family, and Health Network study. Am J Public Health. 2012 Jan;102(1):126-33. doi: 10.2105/AJPH.2011.300323. Epub 2011 Nov 28. PMID 22095360
- [Background] Sabbath EL, Melchior M, Goldberg M, Zins M, Berkman LF. Work and family demands: predictors of all-cause sickness absence in the GAZEL cohort. Eur J Public Health. 2012 Feb;22(1):101-6. doi: 10.1093/eurpub/ckr041. Epub 2011 May 9. PMID 21558153
- [Background] McHale SM, Blocklin MK, Walter KN, Davis KD, Almeida DM, Klein LC. The role of daily activities in youths' stress physiology. J Adolesc Health. 2012 Dec;51(6):623-8. doi: 10.1016/j.jadohealth.2012.03.016. Epub 2012 May 16. PMID 23174474
- [Background] Blocklin MK, Crouter AC, McHale SM. Youth Supervision While Mothers Work: A Daily Diary Study of Maternal Worry. Community Work Fam. 2012;15(2):233-249. doi: 10.1080/13668803.2011.639169. Epub 2011 Dec 2. PMID 23109814
- [Background] Almeida DM, Davis KD. Workplace Flexibility and Daily Stress Processes in Hotel Employees and their Children. Ann Am Acad Pol Soc Sci. 2011 Nov;638(1):123-140. doi: 10.1177/0002716211415608. PMID 23833321
- [Background] Hammer LB, Kossek EE, Anger WK, Bodner T, Zimmerman KL. Clarifying work-family intervention processes: the roles of work-family conflict and family-supportive supervisor behaviors. J Appl Psychol. 2011 Jan;96(1):134-50. doi: 10.1037/a0020927. PMID 20853943
- [Background] Ertel KA, Berkman LF, Buxton OM. Socioeconomic status, occupational characteristics, and sleep duration in African/Caribbean immigrants and US White health care workers. Sleep. 2011 Apr 1;34(4):509-18. doi: 10.1093/sleep/34.4.509. PMID 21461330
- [Background] O'Donnell EM, Ertel KA, Berkman LF. Depressive symptoms in extended-care employees: children, social support, and work-family conditions. Issues Ment Health Nurs. 2011;32(12):752-65. doi: 10.3109/01612840.2011.609958. PMID 22077748
- [Background] Ertel KA, Koenen KC, Berkman LF. Incorporating home demands into models of job strain: findings from the work, family, and health network. J Occup Environ Med. 2008 Nov;50(11):1244-52. doi: 10.1097/JOM.0b013e31818c308d. PMID 19001950
- [Background] Grandner MA, Buxton OM, Jackson N, Sands-Lincoln M, Pandey A, Jean-Louis G. Extreme sleep durations and increased C-reactive protein: effects of sex and ethnoracial group. Sleep. 2013 May 1;36(5):769-779E. doi: 10.5665/sleep.2646. PMID 23633760
- [Background] Marino M, Li Y, Rueschman MN, Winkelman JW, Ellenbogen JM, Solet JM, Dulin H, Berkman LF, Buxton OM. Measuring sleep: accuracy, sensitivity, and specificity of wrist actigraphy compared to polysomnography. Sleep. 2013 Nov 1;36(11):1747-55. doi: 10.5665/sleep.3142. PMID 24179309
- [Background] Kossek EE, Hammer LB, Kelly EL, Moen P. Designing Work, Family & Health Organizational Change Initiatives. Organ Dyn. 2014;43(1):53-63. doi: 10.1016/j.orgdyn.2013.10.007. PMID 24683279
- [Background] Berkman LF, Buxton O, Ertel K, Okechukwu C. Managers' practices related to work-family balance predict employee cardiovascular risk and sleep duration in extended care settings. J Occup Health Psychol. 2010 Jul;15(3):316-29. doi: 10.1037/a0019721. PMID 20604637
- [Background] Kelly EL, Moen P, Tranby E. Changing Workplaces to Reduce Work-Family Conflict: Schedule Control in a White-Collar Organization. Am Sociol Rev. 2011 Apr;76(2):265-290. doi: 10.1177/0003122411400056. PMID 21580799
- [Derived] Berkman LF, Kelly EL, Hammer LB, Mierzwa F, Bodner T, McNamara T, Koga HK, Lee S, Marino M, Klein LC, McDade TW, Hanson G, Moen P, Buxton OM. Employee Cardiometabolic Risk Following a Cluster-Randomized Workplace Intervention From the Work, Family and Health Network, 2009-2013. Am J Public Health. 2023 Dec;113(12):1322-1331. doi: 10.2105/AJPH.2023.307413. PMID 37939328
- [Derived] Hurtado DA, Okechukwu CA, Buxton OM, Hammer L, Hanson GC, Moen P, Klein LC, Berkman LF. Effects on cigarette consumption of a work-family supportive organisational intervention: 6-month results from the work, family and health network study. J Epidemiol Community Health. 2016 Dec;70(12):1155-1161. doi: 10.1136/jech-2015-206953. Epub 2016 May 25. PMID 27225680